CLINICAL TRIAL: NCT00898755
Title: Establishing Continuous Cell Lines and Xenografts From Pediatric Cancers for Biological and Pre-Clinical Therapeutic Studies
Brief Title: Collecting and Storing Tissue From Young Patients With Cancer
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: ABTR04B1; NCI-2009-00326 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000478867; COG-ABTR04B1; ABTR04B1; ABTR04B1 (Other: Children's Oncology Group); ABTR04B1 (Other: CTEP); U10CA098543 (NIH)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2025-05-02 (Actual); Status verified 2025-05

CONDITIONS: Acute Lymphoblastic Leukemia; Acute Myeloid Leukemia; Central Nervous System Neoplasm; Ewing Sarcoma; Germ Cell Tumor; Leukemia; Lymphoma; Malignant Neoplasm; Neuroblastoma; Osteosarcoma; Retinoblastoma; Rhabdoid Tumor; Rhabdomyosarcoma; Soft Tissue Sarcoma
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Central Nervous System Neoplasms; Sarcoma, Ewing; Neoplasms, Germ Cell and Embryonal; Leukemia; Lymphoma; Neoplasms; Neuroblastoma; Osteosarcoma; Retinoblastoma; Rhabdoid Tumor; Rhabdomyosarcoma; Sarcoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Lelftover tissue from diagnostic procedures and/or surgery, blood and bone marrow samples

GROUPS / COHORTS (1):
- Ancillary-Correlative (tissue sample collection): Leftover tissue from diagnostic procedures and/or surgery is cryopreserved and banked. Blood and/or bone marrow are also collected and banked. Cell lines are established and characterized via reverse-transcriptase polymerase chain reaction and/or flow cytometry for biomarkers and by DNA fingerprinting. Markers to be identified may include the following:
  NEUROBLASTOMA: tyrosine hydroxylase, protein gene product (PGP) 9.5, GD2, HLA class I, and HSAN 1.2 antigens EWING FAMILY OF TUMORS: EWS-FLI1, EWS-ERG, and PGP 9.5 RETINOBLASTOMA: interphotoreceptor retinoid-binding protein ACUTE LYMPHOBLASTIC LEUKEMIA: immunophenotype ALVEOLOR RHADOMYOSARCOMA: PAX3-FKHR, PAX7-FKHR, and MyoD1 ALL CELL TYPES: telomerase expression including hTR and hTERTMutations of TP53 gene are detected by flow cytometry and/or immunocytochemistry
  Interventions: Other: Cytology Specimen Collection Procedure; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Other: Cytology Specimen Collection Procedure — Correlative studies
  Other Names: Cytologic Sampling
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This laboratory study is collecting and storing tissue, blood, and bone marrow samples from young patients with cancer. Collecting and storing samples of tissue, blood, and bone marrow from patients with cancer to study in the laboratory may help doctors learn more about changes that may occur in DNA and identify biomarkers related to cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Establish and bank cell lines and/or xenografts from pediatric patients with cancer.

II. Establish continuous cell lines, under carefully controlled conditions, from pediatric patients with cancer.

III. Establish transplantable xenografts in immunocompromised mice from tumor cells that are difficult to establish as continuous cell lines in vitro.

IV. Create a bank of cell lines and generate sufficient vials of cryopreserved cells for distribution to investigators with approved COG biology protocols. V. Characterize cell lines from childhood cancers with respect to DNA short tandem repeat molecular profile as a "fingerprint" of original cell line identity.

VI. Characterize cell lines for the ability for sustained growth in tissue culture and/or as mouse xenografts.

VII. Characterize cell lines for mycoplasma contamination. VIII. Characterize cell lines for expression of molecular makers that confirm the tumor-type of the cell line and the immortal nature of the cells (telomerase) and the expression of molecular markers that may correlate with drug resistance.

OUTLINE: This is a multicenter study.

Specimens are stratified according to disease (acute lymphoblastic leukemia vs acute myeloid leukemia vs lymphoma vs osteogenic sarcoma vs Ewing family of tumors vs rhabdomyosarcoma vs primitive neuroectodermal tumor vs glioma vs astrocytoma vs rhabdoid tumors vs hepatoblastoma vs retinoblastoma vs Wilms tumor vs germ cell tumors vs other diagnoses).

Leftover tissue from diagnostic procedures and/or surgery is cryopreserved and banked. Blood and/or bone marrow are also collected and banked. Cell lines are established and characterized via reverse-transcriptase polymerase chain reaction and/or flow cytometry for biomarkers and by DNA fingerprinting. Markers to be identified may include the following:

NEUROBLASTOMA: tyrosine hydroxylase, protein gene product (PGP) 9.5, GD2, HLA class I, and HSAN 1.2 antigens

EWING FAMILY OF TUMORS: EWS-FLI1, EWS-ERG, and PGP 9.5

RETINOBLASTOMA: interphotoreceptor retinoid-binding protein

ACUTE LYMPHOBLASTIC LEUKEMIA: immunophenotype

ALVEOLOR RHADOMYOSARCOMA: PAX3-FKHR, PAX7-FKHR, and MyoD1

ALL CELL TYPES: telomerase expression including hTR and hTERTMutations of TP53 gene are detected by flow cytometry and/or immunocytochemistry.

No results of these tests are provided to the patient, the patient's physician, or the patient's medical records.

ELIGIBILITY:
Inclusion Criteria:

* All malignant tissues from childhood cancers allowed including the following:

  * Brain tumors (all types)

    * Tissue should be submitted to CNS Committee Resource labs to be forwarded for this study, unless instructed otherwise on the COG web site
  * Ewing family of tumors
  * Rhabdomyosarcomas
  * Other soft tissue sarcomas
  * Osteogenic sarcomas
  * Rhabdoid tumors
  * Neuroblastomas

    * Viable material for cell culture for neuroblastoma is collected via COG-ANBL00B1 and should not be submitted via this study unless the patient cannot be enrolled on COG-ANBL00B1*
  * Retinoblastomas
  * Anaplastic Wilms tumor
  * Germ cell tumors
  * Leukemias/lymphomas

    * Acute myeloid leukemia (AML)

      * Blood samples and bone marrow samples from patients at second relapse and beyond may be submitted for this study
      * Bone marrow samples at diagnosis or first relapse must be submitted to an AML resource lab and will be forwarded for this study at the discretion of the AML Committee
    * Acute lymphoblastic leukemia (ALL)

      * Blood samples may be submitted directly to this study
      * Bone marrow samples must be submitted to an ALL resource lab and will be forwarded for this study at the discretion of the ALL Committee
* Enrolled on a COG therapeutic, biology, or tissue banking protocol that allows collection of tissue for research and submission to a COG-designated resource laboratory

  * Participation in this protocol is not permitted until after tissue requirements for any active COG disease-specific therapeutic, biology, or banking protocols have been satisfied
  * Material may only be submitted for this protocol if tissue is available in excess of that required for satisfying active disease-specific therapeutic and biological protocols
* Patients with diagnosis pending are eligible

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients enrolled on the Children Oncology Group (COG) therapeutic, biologic, or tissue banking protocols that allow collection of tissue for research studies
Sampling Method: Non-Probability Sample
Enrollment: 213 (Estimated)
Dates: Start 2007-03-05 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Establishment and banking of cell lines and/or xenografts from pediatric patients with cancer | Up to 14 years
Establishment of continuous cell lines, under carefully controlled conditions, from pediatric patients with cancer | Up to 14 years
Establishment of transplantable xenografts in immunocompromised mice from tumor cells that are difficult to establish as continuous cell lines in vitro | Up to 14 years
Creation of a bank of cell lines and generation of sufficient vials of cryopreserved cells for distribution to investigators with approved COG biology protocols | Up to 14 years
Characterization of cell lines from childhood cancers with respect to DNA PCR molecular HLA profile as a "fingerprint" of original cell line identity | Up to 14 years
Characterization of cell lines for the ability for sustained growth in tissue culture and/or as mouse xenografts | Up to 14 years
Characterization of cell lines for mycoplasma contamination | Up to 14 years
Characterization of cell lines for expression of molecular makers that confirm the tumor-type of the cell line and the immortal nature of the cells (telomerase) and the expression of molecular markers that may correlate with drug resistance | Up to 14 years

CONTACTS AND LOCATIONS:
Overall Officials: Charles P Reynolds, Principal Investigator — Children's Oncology Group
Locations (68):
- United States (65):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital and Research Center at Oakland, Oakland, California
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Lee Memorial Health System, Fort Myers, Florida
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Tampa General Hospital, Tampa, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Hospital, West Palm Beach, Florida
  - Saint Luke's Mountain States Tumor Institute, Boise, Idaho
  - University of Illinois, Chicago, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Kalamazoo Center for Medical Studies, Kalamazoo, Michigan
  - Columbia Regional, Columbia, Missouri
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Nevada Cancer Research Foundation CCOP, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Albany Medical Center, Albany, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Greenville Cancer Treatment Center, Greenville, South Carolina
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Texas Tech University Health Sciences Center-Amarillo, Amarillo, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - UMC Cancer Center / UMC Health System, Lubbock, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Madigan Army Medical Center, Tacoma, Washington
- Canada (3):
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan